CLINICAL TRIAL: NCT03882229
Title: Middle East MED-EL Observatory Study
Acronym: MEMOS
Status: Recruiting | Type: Observational
Sponsor: MED-EL Elektromedizinische Geräte GesmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: MED-EL_CRD_2018_01
Record Dates: First submitted 2019-03-01; First posted 2019-03-20 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Cochlear Implants
Keywords: Registry; Observational Study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MED-EL CI systems — • Cochlear Implant (CI) and external audio processor

SUMMARY:
In the field of cochlear implant research, there are only few data on long-term observational studies available to gain knowledge on clinical effectiveness. Longitudinal comparisons of data collected in different clinics is challenging due to the heterogeneity in measures and procedure.

This Registry represents a non-interventional systematic collection of clinical data in which prospective data from children and adults are collected as anonymized data sets, derived from original clinical records on appropriately informed subjects. Each subject will be treated as per clinical routine.

The Registry will be implemented through a secure, cloud-based, platform that enables collection of anonymized data at consistent time intervals, thus enabling the comparison of repeated measures over time.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are implanted or will be implanted with a MED-EL CI system.
* Signed written informed consent for data collection for registry purposes.

Exclusion Criteria:

* Lack of compliance with any inclusion criteria.
* Subjects not receiving a MED-EL CI system due to medical or personal reasons after having consented.
* Anything that, in the opinion of the Investigator would place the subject at increased risk or preclude the subject's full compliance with or completion of the registry procedures.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects of any age and gender who are implanted or will be implanted with a MED-EL CI system.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-02-11 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Hearing threshold level | 5 years
  Audiometry testing (unaided)
Quality of hearing - adults | 5 years
  Results from the Hearing Implant Sound Quality Index (HISQUI 19)
Auditory development - children (CAP) | 5 years
  Results from the Categories of Auditory Performance (CAP)
Auditory development - children (SIR) | 5 years
  Results from the Speech Intelligibility Rating (SIR)
Auditory development - children (LEAQ) | 5 years
  Results from the LittlEARS Auditory Questionnaire (LEAQ)

CONTACTS AND LOCATIONS:
Overall Officials: Abdulrahman Ahmed Alsanosi, Prof., Principal Investigator — King Abdullah Ear Specialist Center
Locations (3):
- Hearing and Speech Institute, Cairo, Egypt
- Saudi Arabia (2):
  - King Abdullah Ear Specialist Center (KAESC), Riyadh
  - King Saud Medical City, Riyāḑ

IPD SHARING:
Plan to Share IPD: No